CLINICAL TRIAL: NCT05003622
Title: Multicenter, Open-label, Phase 1 Study Investigating the Safety and Tolerability of Encorafenib Monotherapy in BRAF V600E-mutated Chinese Patients With Advanced Metastatic Solid Tumors
Brief Title: Phase 1 Safety Study of Encorafenib in Chinese Patients With Advanced Metastatic BRAF V600E Mutant Solid Tumors
Acronym: OCEANI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W00090GE102
Record Dates: First submitted 2021-06-24; First posted 2021-08-12 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2022-06

CONDITIONS: BRAF V600E Unresectable or Metastatic Melanoma; BRAF V600E Metastatic NSCLC; Melanoma
Keywords: NSCLC; Melanoma; BRAF V600E mutation
MeSH Terms: conditions — Melanoma | interventions — encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- encorafenib (Experimental): Encorafenib hard capsule will be orally self-administered. A fixed-flat dose of 300 mg (4 x 75 mg) Per Oral (PO) encorafenib will be administered once-daily (QD).
  Interventions: Drug: Encorafenib

INTERVENTIONS:
Drug: Encorafenib — oral capsule
  Other Names: Braftovi®; PF-07263896; W0090; LGX818; ONO-7702

SUMMARY:
This is a phase 1, multicenter, open-label, single-arm study to investigate the safety and tolerability of encorafenib 300 mg once daily (QD) monotherapy in adult Chinese participants with B-RAF Proto-oncogene, Serine/threonine Kinase V600E (BRAF V600E) mutant advanced solid tumors (unresectable metastatic melanoma or metastatic non-small cell lung cancer (NSCLC)), who are BRAF-inhibitor treatment-naïve and have failed the previous therapy(ies) in the metastatic setting or are not eligible to standard therapy. Participants will be eligible for the study based on identification of a BRAF V600E mutation in tumor tissue by a local National Medical Products Administration (NMPA) approved assay obtained prior to screening.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent form (ICF).
2. Chinese male or female with age ≥18 years old at the time of the informed consent.
3. Documented histology- and/or cytology-confirmed metastatic melanoma or non-small cell lung cancer (NSCLC) (i.e. adenocarcinoma, large cell carcinoma, squamous cell carcinoma).
4. Presence of B-RAF Proto-oncogene, Serine/threonine Kinase V600E Mutant (BRAF V600E) mutation as determined by a local laboratory with a National Medical Products Administration (NMPA) approved BRAF test.
5. BRAF inhibitor treatment-naïve participants and having failed the previous therapy(ies) for metastatic disease or are not eligible to standard therapy.
6. At least one tumor lesion as per investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, which has neither been irradiated nor biopsied during the screening period. The irradiated lesion is acceptable only if it is proven as disease progression deemed measurable prior to study.
7. Life expectancy ≥3 months.
8. Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1.
9. Adequate hematologic function at screening and baseline
10. Adequate hepatic function at screening and baseline
11. Adequate renal function at screening and baseline
12. Able to comply with the study protocol as per investigator assessment including oral drug intake, complying scheduled visits, treatment plan, laboratory tests and other study procedures.
13. Women are either postmenopausal for at least 1 year, or are surgically sterile for at least 6 weeks, or women of childbearing potential (WOCBP) must agree to take appropriate precautions to avoid pregnancy.
14. Men must agree not to father child until 90 days after the last dose of study treatment.

Exclusion Criteria:

1. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to encorafenib, or its excipients.
2. For metastatic NSCLC: documented anaplastic lymphoma kinase (ALK) fusion oncogene, ROS1 (c-ros oncogene 1) rearrangement or epidermal growth factor receptor (EGFR) sensitizing or driver mutation.
3. Receipt of anticancer medications or investigational drugs within intervals before the first administration of study treatment.
4. Symptomatic brain metastasis.
5. Leptomeningeal disease.
6. Participant has not recovered to ≤Grade 1 from toxic effects of prior therapy and/or complications from prior surgical treatment before starting study treatment.
7. Current use of prohibited medication ≤1 week prior to start of the study treatment and/or concomitantly.
8. Impairment of gastrointestinal function or disease which may significantly alter the absorption of oral study treatment.
9. Impaired cardiovascular function or clinically significant cardiovascular diseases.
10. Participants with active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) or any other severe viral active infection (e.g. severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] infection).
11. Evidence of active, non-infectious pneumonitis, history of interstitial lung disease that required oral or intravenous glucocorticoid steroids for management.
12. Known history of a positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Testing for HIV must be performed at sites where mandated locally.
13. Participants who have had major surgery (e.g. inpatient procedure with regional or general anesthesia) within 6 weeks prior to start of study treatment.
14. Previous or concurrent malignancy within 2 years of study entry.

    Except:
    1. Bowen's disease.
    2. Cured basal cell or squamous cell skin cancer.
    3. Gleason 6 prostate cancer.
    4. Treated in-situ carcinoma of cervix.
15. Participant's conditions that contraindicates the use of study treatment and may affect interpretation of results or that may render the participant at high risk from treatment complications.
16. Pregnant (confirmed by positive serum beta-human Chorionic Gonadotropin (ß-HCG) test), lactating or breast-feeding women.
17. Is a family member of the Investigator or any associate, colleague, and employee assisting in the conduct of the study (secretary, nurse, technician).
18. Is in a position likely to represent a conflict of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had no fixed duration and participants were expected to be treated until progressive disease. The three enrolled participants were to be treated until death, disease progression.
Groups:
- Encorafenib: Encorafenib hard capsule was orally administered. A fixed-flat dose of 300 mg (4 x 75 mg) Per Oral (PO) encorafenib was administered once-daily (QD).
Period: Overall Study
Arm/Group | Encorafenib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Progressive disease | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 3
Weight [Mean (Standard Deviation); unit: kilograms] | 65.73 (4.87)
Height [Mean (Standard Deviation); unit: centimeters] | 163.07 (5.01)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters squared] | 24.773 (2.437)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The Performance status was assessed by the investigator using the ECOG Performance Status scale Performance status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    Performance Status 0 | 0
    Performance Status 1 | 3
Smoking history [Count of Participants; unit: Participants]
  Never smoked | 0
  Stopped smoking more than or equal to 10 years ago | 0
  Stopped smoking less than 10 years ago | 3
  Smoker | 0
BRAF V600E Mutation Result (Local) [Count of Participants; unit: Participants]
  Positive | 3
  Negative | 0
Diagnosis at study entry [Count of Participants; unit: Participants]
  Metastatic Melanoma | 0
  Metastatic NSCLC | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs) Experienced During Cycle 1
Description: The primary endpoint was the number of patients experiencing dose limiting toxicity (DLT) occurring within the first 28 days of study treatment (Cycle 1). A DLT was defined as any adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness or concomitant medications/therapies resulting in the inability to tolerate at least 75% dose intensity [(administered dose in mg/planned dose in mg) × 100] that satisfied at least one of the prespecified criteria.
Time Frame: At the end of Cycle 1. Each cycle was 28 days.
Population: Dose-determining Set. The Dose-determining set consisted of all evaluable participants from the Safety Analysis Set who either achieved the minimum exposure requirement (i.e., encorafenib dose intensity of 75% in Cycle 1) and had sufficient safety evaluations.
Measure: Number; unit: participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs)
Description: The occurrences of treatment emergent adverse events (TEAEs) graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03, TEAEs leading to dose interruption, reduction and discontinuation, treatment-emergent serious adverse events (SAEs) and deaths were reported. The number of events occurring in the three participants is presented.
Time Frame: Cycle 1 Day 1 through safety follow-up visit (30 days after end of treatment (EOT) visit or 7 days after end EOT visit/last dose if EOT not performed), approximately up to 6 months. Each cycle was 28 days.
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
events
  TEAEs Overall | 53
  TEAEs Related | 17
  TEAEs Grade 3+ | 3
  TEAEs Related Grade 3+ | 2
  Serious TEAE Overall | 3
  Serious TEAE Related | 2
  Serious TEAE Grade 3+ | 2
  Serious TEAE Related Grade 3+ | 1
  Serious TEAE Leading to Death | 0
  TEAE by severity grade Grade 1 | 37
  TEAE by severity grade Grade 2 | 13
  TEAE by severity grade Grade 3 | 3
  TEAE leading to discontinuation of encorafenib regardless of causality Overall | 0
  TEAEs leading to encorafenib dose modification (interruption or reduction) Overall | 6
  TEAEs leading to encorafenib dose modification (interruption or reduction) Related | 4
  TEAEs leading to encorafenib dose modification (interruption or reduction) Grade 3+ | 1
  TEAEs leading to encorafenib dose modification (interruption or reduction) Related Grade 3+ | 1
  TEAEs leading to encorafenib drug interruption Overall | 5
  TEAEs leading to encorafenib drug interruption Related | 4
  TEAEs leading to encorafenib drug interruption Grade 3+ | 1
  TEAEs leading to encorafenib drug interruption Related Grade 3+ | 1
  TEAEs leading to encorafenib dose reduction Overall | 1
  TEAE action taken with encorafenib Dose not Change | 47
  TEAE action taken with encorafenib Dose Reduced | 1
  TEAE action taken with encorafenib Drug Interrupted | 5

3. Secondary Outcome: Notable Change From Baseline of Blood Hematology Parameters: Hemoglobin, Leukocytes, Neutrophils, Platelets, Lymphocytes.
Description: Clinically notable shift from baseline in blood hematology parameters data [Hemoglobin (Low/High); Leukocytes (Low/ High); Neutrophils (Low); Platelets (Low); Lymphocytes (Low/High)] was graded using NCI CTCAE Version 4.03. Clinically notable shift was defined as a worsening from baseline by at least 2 grades, or to grade 3 or above. The number of participants with clinically notable shift from baseline is presented.
Time Frame: Screening (Days -28 to -1), Cycle 1 Day 1 (if not done within 72 hours before the first dose), Cycle 1 Day 15, on Day 1 each subsequent cycle, end of treatment visit 30 day safety follow up visit, approximately up to 6 months. Each cycle was 28 days.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Participants
  Hemoglobin (g/L) (Low) | 0
  Hemoglobin (g/L) (High) | 0
  Platelets (10^9/L) (Low) | 0
  Leukocytes (10^9/L) (Low) | 0
  Leukocytes (10^9/L) (High) | 0
  Lymphocytes (10^9/L) (Low) | 0
  Lymphocytes (10^9/L) (High) | 0
  Neutrophils (10^9/L) (Low) | 0

4. Secondary Outcome: Notable Change From Baseline of Blood Clinical Chemistry Parameters
Description: Clinically notable shift from baseline in blood clinical chemistry parameter values [Phosphate (Low); Alanine Aminotransferase (High); Albumin (Low); Alkaline Phosphatase (High); Aspartate Aminotransferase (High); Bilirubin (High); Calcium Corrected (Low/High); Creatinine (High); Glucose (Low/High); Magnesium (Low/High); Potassium (Low/High); Sodium (Low/High); amylase (high); Gamma Glutamyl Transferase (High); Lipase (High) and Urate (High)] was graded using NCI-CTCAE, Version 4.03. Clinically notable shift was defined as a worsening from baseline by at least 2 grades, or to grade 3 or above. Number of participants with at least one clinically notable shift during study was reported.
Time Frame: as for outcome 3
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Participants
  Albumin (g/L) (Low) | 0
  Alkaline Phosphatase (IU/L) (High) | 0
  Alanine Aminotransferase (IU/L) (High) | 0
  Aspartate Aminotransferase (IU/L) (High) | 0
  Bilirubin (umol/L) (High) | 0
  Calcium Corrected (mmol/L) (Low) | 0
  Calcium Corrected (mmol/L) (High) | 0
  Creatine Kinase (IU/L) (High) | 0
  Creatinine (umol/L) (High) | 0
  Gamma Glutamyl Transferase (IU/L) (High) | 0
  Glucose (mmol/L) (Low) | 0
  Glucose (mmol/L) (High) | 1
  Lipase (IU/L) (High) | 1
  Amylase (IU/L) (High) | 0
  Magnesium (mmol/L) (Low) | 0
  Magnesium (mmol/L) (High) | 0
  Phosphate (mmol/L) (Low) | 0
  Potassium (mmol/L) (Low) | 0
  Potassium (mmol/L) (High) | 0
  Sodium (mmol/L) (Low) | 0
  Sodium (mmol/L) (High) | 0
  Urate (umol/L) (High) | 0

5. Secondary Outcome: Notable Change From Baseline of Coagulation Parameters
Description: The maximum post baseline values of coagulation parameters [activated partial thromboplastin time (seconds) and prothtombin international normalized ratio (INR)]. It was graded using NCI-CTCAE, Version 4.03. The number of participants is presented with their worst NCI-CTCAE grade post-baseline.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL*. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: as for outcome 3
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Participants
  Activated Partial Thromboplastin Time (sec): Grade 0 | 3
  Activated Partial Thromboplastin Time (sec): Grade 1 | 0
  Activated Partial Thromboplastin Time (sec): Grade 2 | 0
  Activated Partial Thromboplastin Time (sec): Grade 3 | 0
  Activated Partial Thromboplastin Time (sec): Grade 4 | 0
  Prothrombin International Normalized Ratio (RATIO): Grade 0 | 2
  Prothrombin International Normalized Ratio (RATIO): Grade 1 | 1
  Prothrombin International Normalized Ratio (RATIO): Grade 2 | 0
  Prothrombin International Normalized Ratio (RATIO): Grade 3 | 0
  Prothrombin International Normalized Ratio (RATIO): Grade 4 | 0

6. Secondary Outcome: Notable Change From Baseline of Dipstick Urinalysis
Description: The appearance of dipstick, at each visit by participant is presented.
Time Frame: Days -28 to -1, Cycle1 Day1 (if not within 72 hours before first dose),Cycle1 Day15,on Day1 each subsequent cycle,end of treatment visit 30 day safety follow up visit, up to 6 months. Additional urinalysis in Cycle 1 Days 8 and 22. Each cycle was 28 days.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Participants
  Baseline: Clear | 3
  Baseline: Cloudy | 0
  Cycle 1 Day 8: Clear | 3
  Cycle 1 Day 8: Cloudy | 0
  Cycle 1 Day 15: Clear | 3
  Cycle 1 Day 15: Cloudy | 0
  Cycle 1 Day 22: Clear | 3
  Cycle 1 Day 22: Cloudy | 0
  Cycle 2 Day 1: Clear | 3
  Cycle 2 Day 1: Cloudy | 0
  Cycle 3 Day 1: Clear | 2
  Cycle 3 Day 1: Cloudy | 1
  Cycle 4 Day 1: Clear | 3
  Cycle 4 Day 1: Cloudy | 0

7. Secondary Outcome: Notable or Abnormal Changes in Vital Signs From Baseline of Vital Sign Examinations.
Description: Clinically notable elevated values: Systolic blood pressure (SBP): ≥ 160 mmHg and an increase ≥ 20 mmHg from baseline; Diastolic blood pressure (DBP): ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline; Heart rate : ≥ 120 beats/min (bpm) with increase from baseline of ≥ 15 bpm; Weight (kg) increase from baseline of ≥ 10%; Body temperature(°C) ≥ 37.5°C). Clinically notable low values: Systolic blood pressure (SBP): ≤ 90 mmHg with decrease from baseline of ≥ 20 mmHg; Diastolic blood pressure (DBP) : ≤ 50 mmHg with decrease from baseline of ≥ 15 mmHg; Heart rate: ≤ 50 bpm with decrease from baseline of ≥ 15 bpm; Weight: ≥ 20% decrease from baseline; Body temperature [°C]: ≤ 36 °C. Number of participants with clinically notable abnormalities in vital signs was reported.
Time Frame: Screening (Days -28 to -1), Cycle 1 Days 1, 8, 15 and 22, Day 1 of each subsequent cycle, the end of treatment visit and the 30-day safety follow-up visit, approximately up to 6 months. Each cycle was 28 days.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Participants
  Clinically notable elevated value: SBP : ≥160 mmHg and an increase ≥ 20 mmHg from baseline | 1
  Clinically notable elevated values: DBP: ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline | 1
  Clinically notable elevated values: Pulse rate: ≥ 120 bpm with increase from baseline of ≥15 bpm | 1
  Clinically notable elevated values: Weight: increase from baseline of ≥ 10% | 0
  Clinically notable elevated values: Body temperature [C]: ≥ 37.5 C | 0
  Clinically notable low values: SBP: ≤ 90 mmHg with decrease from baseline of ≥ 20 mmHg | 0
  Clinically notable low values: DBP: ≤ 50 mmHg with decrease from baseline of ≥ 15 mmHg | 0
  Clinically notable low values: Pulse rate: ≤ 50 bpm with decrease from baseline of ≥ 15 bpm | 0
  Clinically notable low values: Weight: ≥ 20% decrease from baseline | 0
  Clinically notable low values: Body temperature [C]: ≤ 36 C | 1

8. Secondary Outcome: Notable or Abnormal Changes From Baseline of 12-lead Electrocardiograms (ECGs)
Description: 12-lead ECGs were obtained using an internationally recognized 12-lead cardiograph. Clinically notable ECG values: QT [millisecond (ms)] and QT interval (ms) corrected for heart rate using Fridericia's formula (QTcF) intervals (ms): increase from baseline > 30 ms; increase from baseline > 60 ms, new > 450 ms, new > 480 ms, new > 500 ms. Heart rate (beats/min): increase from baseline > 25% to a value > 100 bpm, decrease from baseline > 25% and to a value < 50 bpm. Number of participants with clinically notable values was reported.
Time Frame: Screening (Days -28 to -1), Cycle 1 Day 8, 15 and 22, Day 1 of each subsequent even cycle, and the end of treatment visit, approximately up to 6 months. Each cycle was 28 days.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
Participants
  QT Interval : Increase from baseline > 30 ms | 1
  QT Interval : Increase from baseline > 60 ms | 0
  QT Interval : New > 450 ms | 0
  QT Interval : New > 480 ms | 0
  QT Interval : New > 500 ms | 0
  QTcF Interval : Increase from baseline > 30 ms | 1
  QTcF Interval : Increase from baseline > 60 ms | 0
  QTcF Interval : New > 450 ms | 0
  QTcF Interval : New > 480 ms | 0
  QTcF Interval : New > 500 ms | 0
  Heart rate : Increase from baseline > 25% to a value > 100 bpm | 1
  Heart rate : Decrease from baseline > 25% and to a value < 50 bpm | 0

9. Secondary Outcome: Occurrence of Targeted Treatment Emergent Adverse Events (TEAEs) of Special Interest
Description: Adverse event of special interest (AESI) were as follows: Cutaneous non-squamous cell carcinoma, cutaneous squamous cell carcinoma, melanomas, facial paresis, uveitis-type events, QT prolongation, non-cutaneous malignancies with RAS mutation. Number of participants with at least one event of any AESI is presented.
Time Frame: Cycle 1 Day 1 through safety follow-up visit (30 days after end of treatment [EOT] visit or 7 days after end EOT visit/last dose if EOT not performed), approximately up to 6 months.
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
participants | 0

10. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib: Area Under the Curve (AUC) After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of Encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The Area under the curve of Encorafenib was assessed after single and repeated administrations.
  AUC0-tlast = area under the concentration curve from time 0 to time of last measurable concentration
Time Frame: First day of treatment (Cycle 1 Day 1) and at steady state after 1 month treatment (Cycle 2 Day 1). Each cycle was 28 days.
Population: Pharmacokinetics Set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
h*ng/mL
  Cycle 1 Day 1 AUC0-tlast | 21800 (4620)
  Cycle 2 Day 1 AUC0-tlast | 9550 (1750)

11. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib Metabolite (LHY746): Area Under the Curve (AUC) After Single and Repeated Administration of Encorafenib Metabolite (LHY746)
Description: All enrolled participants (n=3) received at least two doses of Encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The Area under the curve of Encorafenib metabolite (LHY746) was assessed after single and repeated administrations.
  AUC0-tlast = area under the concentration curve from time 0 to time of last measurable concentration
Time Frame: as for outcome 10
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
h*ng/mL
  Cycle 1 Day 1 AUC0-tlast | 2540 (1150)
  Cycle 2 Day 1 AUC0-tlast | 6020 (3330)

12. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib: Maximum Concentration (Cmax) After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The Maximum Concentration of encorafenib was assessed after single and repeated administrations.
Time Frame: as for outcome 10
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
(ng/mL)
  Cycle 1 Day 1 Cmax | 5590 (351)
  Cycle 2 Day 1 Cmax | 3630 (1750)

13. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib Metabolite (LHY746): Maximum Concentration (Cmax) After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The Maximum Concentration of encorafenib metabolite (LHY746) was assessed after single and repeated administrations.
Time Frame: as for outcome 10
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
ng/mL
  Cycle 1 Day 1 Cmax | 610 (247)
  Cycle 2 Day 1 Cmax | 1420 (582)

14. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib: Minimum Concentration (Cmin) After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The Minimum concentration of encorafenib was assessed after single and repeated administrations.
Time Frame: as for outcome 10
Population: pharmacokinetic set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
ng/mL
  Cycle 1 Day 1 Cmin | NA (NA) — values were below the limit of quantification
  Cycle 2 Day 1 Cmin | 10.5 (6.76)

15. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib Metabolite (LHY746): Minimum Concentration (Cmin) After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The Minimum concentration of encorafenib metabolite (LHY746) was assessed after single and repeated administrations.
Time Frame: as for outcome 10
Population: Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
ng/mL
  Cycle 1 Day 1 Cmin | NA (NA) — Values were below the limit of quantification
  Cycle 2 Day 1 Cmin | 109 (91.7)

16. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib: Time Taken to Reach Maximum Concentration (Tmax) After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The time taken to reach maximum concentration of Encorafenib was assessed after single and repeated administrations.
Time Frame: as for outcome 10
Population: Pharmacokinetic Set
Measure: Median (Full Range); unit: hours
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
hours
  Cycle 1 Day 1 tmax | 2.00 [1.00 to 4.03]
  Cycle 2 Day 1 tmax | 1.00 [1.00 to 4.00]

17. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib Metabolite (LHY746): Time Taken to Reach Maximum Concentration (Tmax) After Single and Repeated Administration of Encorafenib Metabolite (LHY746)
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The time taken to reach maximum concentration of Encorafenib Metabolite (LHY746) was assessed after single and repeated administrations.
Time Frame: as for outcome 10
Population: Pharmacokinetic Set
Measure: Median (Full Range); unit: hours
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
hours
  Cycle 1 Day 1 tmax | 5.98 [5.92 to 6.00]
  Cycle 2 Day 1 tmax | 2.00 [1.97 to 4.00]

18. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib: ARAUC After Single and Repeated Administration of Encorafenib
Description: All enrolled participants (n=3) received at least two doses of Encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The ARAUC of Encorafenib was assessed after single and repeated administrations.
  ARAUC = Observed accumulation ratio based on AUC0-6
Time Frame: at steady state after 1 month treatment (Cycle 2 Day 1). Each cycle was 28 days.
Population: Pharmacokinetics Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
ratio | 0.440 (40.2)

19. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib Metabolite (LHY746): ARAUC After Single and Repeated Administration of Encorafenib Metabolite (LHY746)
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The ARAUC of encorafenib metabolite (LHY746) was assessed after single and repeated administrations.
  ARAUC = Observed accumulation ratio based on AUC0-6
Time Frame: at steady state after 1 month treatment (Cycle 2 Day 1). Each cycle was 28 days.
Population: Pharmacokinetics Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
ratio | 2.27 (18.2)

20. Secondary Outcome: Plasma Pharmacokinetics (PK) of Encorafenib Metabolite (LHY746): MRAUC After Single and Repeated Administration of Encorafenib Metabolite (LHY746)
Description: All enrolled participants (n=3) received at least two doses of encorafenib, did all the planned PK blood collection with associated bioanalytical results and were therefore included in the PK Set. The MRAUC of encorafenib metabolite (LHY746) was assessed after single and repeated administrations.
  MRAUC = Metabolite Parent ratio based on AUC0-6
Time Frame: as for outcome 10
Population: Pharmacokinetics Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Encorafenib
Number analyzed (Participants) | 3
ratio
  Cycle 1 Day 1 | 0.141 (53.1)
  Cycle 2 Day 1 | 0.730 (41.3)

ADVERSE EVENTS:
Time Frame: All adverse events were collected for approximately 6 months, from when the participant first provided informed consent until the 30-day safety follow-up visit.
Arm/Group | Encorafenib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Encorafenib (N=3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Encorafenib (N=3)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Neutrophil count increased (Investigations) | 3 (5)
Blood cholesterol increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Coagulation time prolonged (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
Urinary occult blood (Investigations) | 1 (2)
White blood cell count increased (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Subcutaneous abscess (Infections and infestations) | 1 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for the release of SAE of study drug/product defects of the institution, institution and/or investigator shall promptly notify sponsor of the content to be released before releasing other research information and obtain sponsor's consent. If there is no response from sponsor within 60 working days after issuance or specific reason for disagreement and modification suggestions are not listed in the response, it shall be deemed that sponsor agrees.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT05003622/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT05003622/SAP_001.pdf